CLINICAL TRIAL: NCT00042237
Title: Treatment of Women With Depression and Sexual Abuse
Brief Title: Treatment of Depressed Women Who Have Been Sexually Abused
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21MH060216 (NIH); R21MH060216 (NIH); DSIR AT-AS
Record Dates: First submitted 2002-07-24; First posted 2002-07-26 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Depression
Keywords: Child Abuse, Sexual
MeSH Terms: conditions — Depression; Coitus | interventions — Schema Therapy

INTERVENTIONS:
Behavioral: Schema Therapy

SUMMARY:
The purpose of this study is to compare Schema-Focused Therapy plus antidepressant medication and antidepressant medication alone for the treatment of major depression in women with a history of childhood sexual abuse.

DETAILED DESCRIPTION:
Schema-Focused (SF) Therapy is an extension of cognitive therapy that was developed to address the treatment needs of patients with long-standing mental disorders. SF therapy focuses on early maladaptive schemas (EMS): broad, pervasive themes regarding oneself and one's relationship with others, developed during childhood and elaborated throughout one's lifetime, which are dysfunctional to a significant degree. SF Therapy involves the identification of the particular EMS that is most relevant for each patient and attempts to modify the relevant schemas by altering the distorted views of self and others.

Participants are assessed pretreatment, after 12 weeks, posttreatment, and 3 and 6 months posttreatment. The severity of depressive symptomatology is measured and a self-report Beck Depression Inventory is administered. At the end of the study and at the follow-up intervals, participants are given the Longitudinal Interval Follow-up Evaluation, an instrument that assesses the severity of depression and dysthymia symptoms.

ELIGIBILITY:
Inclusion criteria:

* Major depression
* History of childhood sexual abuse

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2001-09

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States